CLINICAL TRIAL: NCT03062943
Title: A Pilot Study of Nintedanib for LymphAngioleioMyomatosis (LAM)
Brief Title: A Study of Nintedanib for LymphAngioleioMyomatosis (LAM)
Acronym: LAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Multimedica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IISS LAM
Record Dates: First submitted 2016-10-07; First posted 2017-02-24 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Lymphangioleiomyomatosis
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nintedanib 150mg BID (Experimental): nintedanib soft gelatine capsules Dose: 150 mg bid Mode of admin. : Oral Duration of treatment: 1 year Duration of follow-up: 12 months after treatment discontinuation
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib
  Other Names: OFEV

SUMMARY:
This trial is conducted locally. The aim of this trial is assess the efficacy and a favorable benefit-risk ratio for nintedanib in the treatment of LAM at the dose of 150 mg bid

DETAILED DESCRIPTION:
There is a high unmet medical need for efficacious and safe treatment of LAM, to halt lung function decline, improve patient-reported outcome, reduce size of angiomyolipomas and ultimately decrease mortality. Guidelines recommend participation in research trials if possible.

To date, therapeutic options include mTOR inhibitors sirolimus and everolimus. Among these, sirolimus, has been approved by FDA based on a clinical trial which showed a stabilization of lung function expressed as FEV1 during the 12 month treatment period. Thus the stabilization of lung function appears to require continuous exposure to the drug. Sirolimus is associated with an increased frequency of adverse events like mucositis, gastrointestinal events, hypercholesterolemia, acneiform rash, and swelling in the lower extremities.

Nintedanib was shown to dose-dependently inhibit PDGFR phosphorylation and subsequent signaling via protein kinase B (Akt) and extracellular signal-regulated kinase (ERK) 1/2 in lung tissue from mice. Akt and ERK 2 can both phosphorylate tuberin resulting in inactivation of hamartin-tuberin complex and consequent activation of mTOR .

It has been demonstrated that platelet-derived growth factor β receptor (PDGFRβ) is present and active in human and murine TSC lesions. Thus, an inhibition of PDGFR may be effective in LAM. Moreover, the inhibition of VEGF, PDGF and FGF signaling pathways reduces tumor angiogenesis in lung. As angiogenesis and lymphangiogenesis are mechanisms involved in dissemination of LAM cells, potential inhibition of angiogenesis by nintedanib may contribute to prevent disease progression in LAM.

Therefore, a non-randomized, efficacy, safety, and tolerability trial of nintedanib in sporadic and TSC-associated LAM is proposed.

The objective of the trial is to assess the efficacy and a favorable benefit-risk ratio for nintedanib in the treatment of LAM at the dose of 150 mg bid.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent for participating to trial.
* Patient aged ≥ 18 years at visit 1.
* Sporadic or TSC associated LAM, classified as ''definite'' by the European Respiratory Society criteria and /or serum VEGFD level >/= 800 mg/ml, and evidence of a 10% deterioration in FEV1 and /or loss of 80 ml of FEV1 or more in the last year (post bronchodilator). Also LAM patients with proven side effects and/or toxicities/ contraindications to sirolimus therapy will be eligible for this study.

Exclusion Criteria:

Laboratory parameters have to satisfy entry criteria as shown below:

* Laboratory parameters (screening)

  * AST, ALT > 1.5 x ULN
  * Bilirubin > 1.5 x ULN
* Positivity for HIV or Hepatitis.
* Chylous effusions.
* Relapsing pneumothorax.
* Angiomyolipoma > 5 cm.
* Treatment with mTOR inhibitors in the last month.
* Patient eligible for Lung Transplantation.
* Hormone therapy.
* Patients are excluded if they are post lung transplant or had previously been diagnosed with a pneumothorax, chylous effusion, bleeding angiomyolipoma within the previous 6 months.
* Current smokers.
* Other diseases:

  * Cardiac disease.
  * Myocardial infarction within 6 months of visit 2.
  * Unstable angina within 1 month of visit 2.
* Bleeding Risk:

  * Known genetic predisposition to bleeding.
* Patients who require fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, heparin, NOA) or high dose antiplatelet therapy2.
* History of haemorrhagic central nervous system (CNS) event within 12 months prior to visit 1.
* History of haemoptysis or haematuria, active gastro-intestinal bleeding or ulcers and/or major injury or surgery within 3 months prior to visit 1.
* International normalised ratio (INR) > 2 at visit 1.
* Prothrombin time (PT) and partial thromboplastin time (PTT) > 150% of institutional ULN at visit 1.
* Planned major surgery during the trial participation, including lung transplantation, major abdominal or major intestinal surgery.
* History of thrombotic event (including stroke and transient ischemic attack) within 12 months of visit 1.
* History of end-stage renal disease requiring dialysis.
* Alcohol or drug abuse which in the opinion of the treating physician would interfere with treatment.
* Pts that cannot perform PFT and cannot give informed consent.
* Known hypersensitivity to the trial drug or its components.
* Other disease that may interfere with testing procedures or in the judgement of the Investigator may interfere with trial participation or may put the patient at risk when participating in this trial.

General Exclusion Criteria:

* Previous treatment with nintedanib.
* Other investigational therapy (participation in research trial) received within 8 weeks of visit.
* Thoracic, abdominal, gynecological, neurologic surgical procedures planned to occur during trial period.
* Pregnant women or women who are breast feeding or of child bearing potential not using two effective methods of birth control (one barrier and one highly effective non-barrier) for at least 1 month prior to enrolment (and until 3 months after treatment end).
* Female patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation, or postmenopausal for at least two years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
FEV1 rate decline | up to 12 months
  Change in FEV1 (Force Expiratory Volume in 1 second) in milliliters per month. The FEV1 slope will be calculated at baseline and at 3, 6, 9 and up to 12 months during the treatment phase.

SECONDARY OUTCOMES:
Safety and Tolerability in terms of AEs, particularly for liver function and level of hepatic enzymes. | up to 12 months
  Safety and Tolerability profile: assessment of any AEs, increased levels of hepatic enzymes, kidney and gastrointestinal tract functionality. All the adverse events will be classified depending of time of occurency: treatment emergent adverse events if they occur after the first dose of study medication up to a period of 28 days or alternatively as either to the screening or post treatment, or post study phase, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio A Harari, MD, Principal Investigator — MultiMedica - San Giuseppe Hospital
Locations (1):
- Pneumology unit, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma L, Chen Z, Erdjument-Bromage H, Tempst P, Pandolfi PP. Phosphorylation and functional inactivation of TSC2 by Erk implications for tuberous sclerosis and cancer pathogenesis. Cell. 2005 Apr 22;121(2):179-93. doi: 10.1016/j.cell.2005.02.031. PMID 15851026
- [Result] Wollin L, Maillet I, Quesniaux V, Holweg A, Ryffel B. Antifibrotic and anti-inflammatory activity of the tyrosine kinase inhibitor nintedanib in experimental models of lung fibrosis. J Pharmacol Exp Ther. 2014 May;349(2):209-20. doi: 10.1124/jpet.113.208223. Epub 2014 Feb 20. PMID 24556663
- [Result] Inoki K, Li Y, Zhu T, Wu J, Guan KL. TSC2 is phosphorylated and inhibited by Akt and suppresses mTOR signalling. Nat Cell Biol. 2002 Sep;4(9):648-57. doi: 10.1038/ncb839. PMID 12172553
- [Result] Crino L, Metro G. Therapeutic options targeting angiogenesis in nonsmall cell lung cancer. Eur Respir Rev. 2014 Mar 1;23(131):79-91. doi: 10.1183/09059180.00008913. PMID 24591665
- [Derived] Harari S, Elia D, Caminati A, Geginat J, Luisi F, Pelosi G, Specchia C, Torre O, Trevisan R, Vasco C, Zompatori M, Cassandro R. Nintedanib for patients with lymphangioleiomyomatosis: a phase 2, open-label, single-arm study. Lancet Respir Med. 2024 Dec;12(12):967-974. doi: 10.1016/S2213-2600(24)00217-0. Epub 2024 Oct 25. PMID 39489895